CLINICAL TRIAL: NCT00580840
Title: A Phase IIIb Open-label run-in Double-blind, Placebo Controlled, Randomized Study to Evaluate the Safety/Efficacy of Certolizumab Pegol Administered Concomitantly With Stable-dose Methotrexate in Patients With Active Rheumatoid Arthritis.
Brief Title: Dosing Flexibility Study in Patients With Rheumatoid Arthritis
Acronym: DoseFlex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C87077; 2007-005288-86 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Results first posted 2012-03-19 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2012-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Joint Disease; Arthritis; Certolizumab pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid; Joint Diseases; Arthritis | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Certolizumab pegol 400 mg and placebo (Active Comparator): 400 mg certolizumab pegol given every 4 weeks and placebo given every 4 weeks given as two injections (alternating injections every two weeks)
  Interventions: Drug: Certolizumab pegol; Other: Placebo
- Certolizumab pegol 200 mg and placebo (Experimental): 200 mg certolizumab pegol and placebo administered every 2 weeks (one injection of each)
  Interventions: Drug: Certolizumab pegol; Other: Placebo
- Placebo (Placebo Comparator): Placebo administered as two injections every 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Certolizumab pegol — 400 mg certolizumab pegol given every 4 weeks and placebo given every 4 weeks given as two injections (alternating injections every two weeks)
  Other Names: CZP; Cimzia
  Arms: Certolizumab pegol 400 mg and placebo
Drug: Certolizumab pegol — 200 mg certolizumab pegol and placebo administered every 2 weeks (one injection of each)
  Other Names: CZP; Cimzia
  Arms: Certolizumab pegol 200 mg and placebo
Other: Placebo — placebo (saline) administered as two injections every 2 weeks

SUMMARY:
During the run-in period, CZP will be administered at 400 mg (2 injections) at Wks 0, 2, and 4 and 200 mg with placebo (1 injection placebo, 1 injection CZP) at Wks 6, 8, 10, 12, 14 and 16. At Wk 18 patients will be grouped as responders or non-responders based on results of the ACR20 at Week 16.

DETAILED DESCRIPTION:
Subjects with a stable methotrexate (MTX) dose enter the run-in period in which certolizumab pegol (CZP) will be administered at a dose of 400 mg (2 injections) at Weeks 0, 2, and 4 and at a dose of 200 mg with placebo (1 injection placebo, 1 injection CZP) at Weeks 6, 8, 10, 12, 14 and 16. The dose of MTX should be stable for at least 2 months prior to the Baseline visit and will remain stable throughout the trial, unless there is a need to reduce the dose for reasons of toxicity.

At the Week 18 visit, subjects who were ACR20 (American College of Rheumatology 20% Improvement) responders at Week 16 will be randomized in a double-blinded way to receive either 400 mg CZP given every 4 weeks and placebo given every 4 weeks given as two injections (alternating CZP and placebo every two weeks) plus MTX, 200 mg CZP and placebo administered every 2 weeks (one injection of each) plus MTX, or Placebo administered as two injections every 2 weeks plus MTX. Non-responders will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with established adult rheumatoid arthritis currently on Methotrexate for at least 3 months

Exclusion Criteria:

* All concomitant diseases or pathological conditions that could interfere and impact the assessment of the study treatment
* Previous clinical trials participation and previous biological therapy that could interfere with the results of the present clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2007-12; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493
Locations (66):
- United States (50):
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Gilbert, Arizona
  - Paradise Valley, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Huntington Beach, California
  - La Jolla, California
  - Los Angeles, California
  - Palm Desert, California
  - Sacramento, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Aventura, Florida
  - Clearwater, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Melbourne, Florida
  - Sarasota, Florida
  - Bogart, Georgia
  - Morton Grove, Illinois
  - Vernon Hills, Illinois
  - Lexington, Kentucky
  - Portland, Maine
  - Haverhill, Massachusetts
  - Pittsfield, Massachusetts
  - Worcester, Massachusetts
  - Rochester, Minnesota
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Albany, New York
  - Mineola, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Monroe, North Carolina
  - Wilmington, North Carolina
  - Cleveland, Ohio
  - Perrysburg, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Simpsonville, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Tyler, Texas
  - Vancouver, Washington
- Canada (7):
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Burlington, Ontario
  - Saint Catherine's, Ontario
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
- France (9):
  - Bobigny
  - Le Havre
  - Lille
  - Limoges
  - Montivilliers
  - Nice
  - Paris
  - Perpigan
  - Saint-Etienne

REFERENCES:
- [Derived] Furst DE, Shaikh SA, Greenwald M, Bennett B, Davies O, Luijtens K, Staelens F, Koetse W, Bertin P. Two dosing regimens of certolizumab pegol in patients with active rheumatoid arthritis. Arthritis Care Res (Hoboken). 2015 Feb;67(2):151-60. doi: 10.1002/acr.22496. PMID 25302624
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in December 2007 with subjects from Canada, France, and United States. The primary completion date occurred in December 2010, with study completion in March 2011.
Groups:
- Overall: Overall for the Run-in period includes all 333 subjects that entered the study. Overall for the Double-blind period includes all 209 subjects that completed the Run-in period.
- CZP 400 mg and PLO + MTX: Certolizumab Pegol (CZP) 400 mg and Placebo (PLO) + Methotrexate (MTX)
- CZP 200 mg and PLO + MTX: Certolizumab Pegol (CZP) 200 mg and Placebo (PLO) + Methotrexate (MTX)
- PLO + MTX: Placebo (PTO) + Methotrexate (MTX)
Period: Run-in
Arm/Group | Overall | CZP 400 mg and PLO + MTX | CZP 200 mg and PLO + MTX | PLO + MTX
Started | 333 (620 subjects were screened for the study with 333 being enrolled.) | 0 | 0 | 0
Completed | 209 (Of the 209 randomized participants, 208 are in the Full Analysis Set (FAS).) | 0 | 0 | 0
Not Completed | 124 | 0 | 0 | 0
Not completed — Adverse Event | 17 | 0 | 0 | 0
Not completed — Lack of Efficacy | 93 | 0 | 0 | 0
Not completed — Loss of Efficacy | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0
Not completed — Other: Per Sponsor Request | 2 | 0 | 0 | 0
Not completed — Other: Did Not Meet Joint Count Criteria | 1 | 0 | 0 | 0
Not completed — Other: Exclusionary Lab Value | 1 | 0 | 0 | 0
Period: Double-Blind
Arm/Group | Overall | CZP 400 mg and PLO + MTX | CZP 200 mg and PLO + MTX | PLO + MTX
Started | 0 | 70 | 70 | 69
Completed | 0 | 63 | 61 | 54
Not Completed | 0 | 7 | 9 | 15
Not completed — Adverse Event | 0 | 3 | 4 | 1
Not completed — Loss of Efficacy | 0 | 1 | 2 | 10
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2
Not completed — Other: Discontinued Methotrexate | 0 | 1 | 0 | 0
Not completed — Other: Forbidden Medication | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Run-in Overall: Overall includes all 333 subjects that entered the Run-in period of the study
Arm/Group | Run-in Overall
Number analyzed (Participants) | 333
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 264
  >=65 years | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (12.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253
  Male | 80
Region of Enrollment [Number; unit: participants]
  France | 7
  United States | 306
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of ACR20 (American College of Rheumatology 20% Improvement) Responders at Week 34 in Patients Randomized at Week 18
Description: ACR20 responders are subjects with at least 20% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 208 subjects (69 400 mg CZP, 70 200 mg CZP, 69 placebo) are included in this analysis which uses Non-Response Imputation (NRI).
Measure: Number; unit: percentage of subjects
Groups:
- Certolizumab Pegol 400 mg and Placebo + Methotrexate: 400 mg certolizumab pegol given every 4 weeks and placebo given every 4 weeks given as two injections (alternating injections every two weeks) plus a subject specific dose of methotrexate
- Certolizumab Pegol 200 mg and Placebo + Methotrexate: 200 mg certolizumab pegol and placebo administered every 2 weeks (one injection of each) plus a subject specific dose of methotrexate
- Placebo + Methotrexate: Placebo administered as two injections every 2 weeks plus a subject specific dose of methotrexate
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 69
percentage of subjects | 65.2 | 67.1 | 44.9

2. Secondary Outcome: Percentage of ACR20 (American College of Rheumatology 20% Improvement) Responders at Week 16 in All Patients
Description: as for outcome 1
Time Frame: Baseline, Week 16
Population: Since Non-Response Imputation (NRI) was used, all 333 subjects in the run-in period are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Run-in Overall
Number analyzed (Participants) | 333
percentage of subjects | 61.3

3. Secondary Outcome: Percentage of ACR50 (American College of Rheumatology 50% Improvement) Responders at Week 16 in All Patients
Description: ACR50 responders are subjects with at least 50% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Baseline, Week 16
Population: Since Non-Response Imputation (NRI) was used, all 333 subjects in the run-in period are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Run-in Overall
Number analyzed (Participants) | 333
percentage of subjects | 37.8

4. Secondary Outcome: Percentage of ACR70 (American College of Rheumatology 70% Improvement) Responders at Week 16 in All Patients
Description: ACR70 responders are subjects with at least 70% improvement from Baseline for tender joint count (TJC), swollen joint count (SJC), and at least 3 of the 5 remaining core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein (CRP), 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale. Missing values were imputed using Non-Responder Imputation (NRI)
Time Frame: Baseline, Week 16
Population: Since Non-Response Imputation (NRI) was used, all 333 subjects in the run-in period are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Run-in Overall
Number analyzed (Participants) | 333
percentage of subjects | 16.2

5. Secondary Outcome: Change From Baseline in DAS28 (Disease Activity Score-28 Items) at Week 16 in All Patients
Description: DAS28-ESR is calculated using the tender joint count (TJC), swollen joint count (SJC) erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
  < 2.6 Remission,
  > = 2.6 - < =3.2 Low, > 3.2 - < = 5.1 Moderate, > 5.1 High
Time Frame: Baseline, Week 16
Population: Of the 333 subjects in the Run-in period, 325 are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Run-in Overall
Number analyzed (Participants) | 325
units on a scale | -2.3 (1.3)

6. Secondary Outcome: Change From Baseline in SDAI (Simplified Disease Activity Index) at Week 16 in All Patients
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
  <= 3.3 Remission, > 3.3 - <= 11 Low, > 11 - <= 26 Moderate, > 26 High
Time Frame: Baseline, Week 16
Population: Of the 333 subjects in the Run-in period, 326 are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Run-in Overall
Number analyzed (Participants) | 326
units on a scale | -24.1 (13.5)

7. Secondary Outcome: Change From Baseline in CDAI (Clinical Disease Activity Index) at Week 16 in All Patients
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
  The range for the CDAI is 0 - 76 with a negative change in CDAI score indicating an improvement in disease activity and a positive change in score indicating a worsening of disease activity.
Time Frame: Baseline, Week 16
Population: Of the 333 subjects in the Run-in period, 328 are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Run-in Overall
Number analyzed (Participants) | 328
units on a scale | -23.3 (13.2)

8. Secondary Outcome: DAS28 (Disease Activity Score-28 Items) Remission (DAS28 <2.6) at Week 16 in All Patients
Description: DAS28-ESR is calculated using the tender joint count (TJC), swollen joint count (SJC) erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI).
  < 2.6 (Remission),
  > = 2.6 - < =3.2 Low, > 3.2 - < = 5.1 Moderate, > 5.1 High
Time Frame: Week 16
Population: Since Non-Response Imputation (NRI) was used, all 333 subjects in the run-in period are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Run-in Overall
Number analyzed (Participants) | 333
percentage of subjects | 17.7

9. Secondary Outcome: SDAI (Simplified Disease Activity Index) Remission (SDAI ≤3.3) at Week 16 in All Patients
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI).
  <= 3.3 (Remission), > 3.3 - <= 11 Low, > 11 - <= 26 Moderate, > 26 High
Time Frame: Week 16
Population: Since Non-Response Imputation (NRI) was used, all 333 subjects in the run-in period are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Run-in Overall
Number analyzed (Participants) | 333
percentage of subjects | 15.9

10. Secondary Outcome: CDAI (Clinical Disease Activity Index) Remission (CDAI ≤2.8) at Week 16 in All Patients
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. Missing values were imputed using Non-Responder Imputation (NRI).
  The range for the CDAI is 0 - 76 with a lower CDAI score indicating approvement in activity and a higher score indicating a decline activity.
Time Frame: Week 16
Population: Since Non-Response Imputation (NRI) was used, all 333 subjects in the run-in period are included in this analysis
Measure: Number; unit: percentage of subjects
Arm/Group | Run-in Overall
Number analyzed (Participants) | 333
percentage of subjects | 17.1

11. Secondary Outcome: Ratio From Baseline in CRP (C-reactive Protein) Level at Week 16 in All Patients
Description: Ratio is defined as the CRP value at Week 16 divided by the CRP value at Baseline. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 16
Population: Of the 333 subjects in the Run-in period, 330 are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Run-in Overall
Number analyzed (Participants) | 330
Ratio | 0.5 (122.6)

12. Secondary Outcome: Change From Baseline in HAQ-DI (Health Assessment Questionnaire-Disability Index) Score at Week 16 in All Patients
Description: HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living actives (using 20 questions). Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Thus, the mean also has a range from 0-3. Change from baseline is computed as the value at Week 16 minus the baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 16
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Run-in Overall
Number analyzed (Participants) | 330
units on a scale | -0.5 (0.6)

13. Secondary Outcome: Percentage of ACR50 (American College of Rheumatology 50% Improvement) Responders at Week 34 in Patients Randomized at Week 18
Description: as for outcome 3
Time Frame: Baseline, Week 34
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 69
percentage of subjects | 52.2 | 50.0 | 30.4

14. Secondary Outcome: Percentage of ACR70 (American College of Rheumatology 70% Improvement) Responders at Week 34 in Patients Randomized at Week 18
Description: as for outcome 4
Time Frame: Baseline, Week 34
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 69
percentage of subjects | 37.7 | 30.0 | 15.9

15. Secondary Outcome: Change From Baseline in DAS28 (Disease Activity Score-28 Items) at Week 34 in Patients Randomized at Week 18
Description: DAS28-ESR is calculated using the tender joint count (TJC), swollen joint count (SJC) erythrocyte sedimentation rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in mm) using the following formula: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x Global Assessment of Arthritis where 28 joints are examined and a lower score indicates less disease activity. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward.
  < 2.6 Remission,
  > = 2.6 - < =3.2 Low, > 3.2 - < = 5.1 Moderate, > 5.1 High
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 204 subjects (69 400 mg CZP, 68 200 mg CZP, 67 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 68 | 67
units on a scale | -3.04 (0.163) | -2.83 (0.164) | -1.65 (0.166)

16. Secondary Outcome: Change From Baseline in SDAI (Simplified Disease Activity Index) at Week 34 in Patients Randomized at Week 18
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), C-reactive protein (CRP in mg/dL), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
  <= 3.3 Remission, > 3.3 - <= 11 Low, > 11 - <= 26 Moderate, > 26 High
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 205 subjects (68 400 mg CZP, 70 200 mg CZP, 67 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 68 | 70 | 67
units on a scale | -30.46 (1.554) | -28.15 (1.532) | -17.35 (1.571)

17. Secondary Outcome: Change From Baseline in CDAI (Clinical Disease Activity Index) at Week 34 in Patients Randomized at Week 18
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm), and Investigator's Global Assessment of Disease Activity - Visual Analog Scale (VAS in cm). 28 joints are examined where a lower score indicates less disease activity. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score. Range for CDAI is 0-76 with a lower CDAI score reflects approvement in activity and a higher score reflects a decline.
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 206 subjects (69 400 mg CZP, 70 200 mg CZP, 67 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 67
units on a scale | -29.06 (1.509) | -27.14 (1.498) | -17.03 (1.536)

18. Secondary Outcome: DAS28 (Disease Activity Score-28 Items) Remission (DAS28 <2.6) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 8
Time Frame: Week 34
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 69
percentage of subjects | 29.0 | 18.6 | 5.8

19. Secondary Outcome: SDAI (Simplified Disease Activity Index) Remission (SDAI ≤3.3) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 9
Time Frame: Week 34
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 69
percentage of subjects | 29.0 | 17.1 | 13.0

20. Secondary Outcome: CDAI (Clinical Disease Activity Index) Remission (CDAI ≤2.8) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 10
Time Frame: Week 34
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 69
percentage of subjects | 27.5 | 21.4 | 15.9

21. Secondary Outcome: Ratio From Baseline in CRP (C-reactive Protein) Level at Week 34 in Patients Randomized at Week 18
Description: Ratio is defined as the CRP value at Week 34 divided by the CRP value at Baseline. This analysis was carried out using the Last Observation Carried Forward (LOCF) method with an ANCOVA model on observed log transformed data with factors treatment and log transformed Baseline CRP level. The number presented is the geometric least squares mean with it's 95% confidence interval.
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 207 subjects (69 400 mg CZP, 70 200 mg CZP, 68 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 68
Ratio | 0.44 [0.36 to 0.53] | 0.48 [0.40 to 0.58] | 0.82 [0.68 to 0.99]

22. Secondary Outcome: Change From Baseline in HAQ-DI (Health Assessment Questionnaire-Disability Index) Score at Week 34 in Patients Randomized at Week 18
Description: HAQ-DI is derived based on the mean of individual scores in 8 categories of daily living actives (using 20 questions). Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). Thus, the mean also has a range from 0-3. Change from baseline is computed as the value at Week 34 minus the baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 68
units on a scale | -0.64 (0.060) | -0.72 (0.060) | -0.38 (0.061)

23. Secondary Outcome: Change From Baseline in Fatigue Assessment Scale (FAS) at Week 34 in Patients Randomized at Week 18
Description: Change from Baseline in Fatigue Assessment scale (0 to 10, 0 is "No Fatigue" and 10 is "Fatigue as bad as you can imagine") is computed as the value at Week 34 minus the Baseline value. A negative value in change from baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 16
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 68 | 70 | 67
units on a scale | -2.39 (0.261) | -3.03 (0.258) | -1.33 (0.264)

24. Secondary Outcome: Change From Baseline in Physical Functioning (Short Form 36-item Health Survey Domain) at Week 34 in Patients Randomized at Week 18
Description: There are 8 SF-36 domain scores: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, each ranging from 0 to 100, with higher scores indicating better health. A larger positive value in change from Baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 68
units on a scale | 8.39 (1.080) | 9.07 (1.076) | 4.09 (1.086)

25. Secondary Outcome: Change From Baseline in Role Physical (Short Form 36-item Health Survey Domain) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 24
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 206 subjects (69 400 mg CZP, 69 200 mg CZP, 68 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 69 | 68
units on a scale | 9.80 (1.095) | 11.06 (1.097) | 7.14 (1.099)

26. Secondary Outcome: Change From Baseline in Bodily Pain (Short Form 36-item Health Survey Domain) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 24
Time Frame: Baseline, Week 34
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 69 | 68
units on a scale | 12.95 (1.042) | 11.28 (1.044) | 6.12 (1.047)

27. Secondary Outcome: Change From Baseline in General Health (Short Form 36-item Health Survey Domain) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 24
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 205 subjects (68 400 mg CZP, 69 200 mg CZP, 68 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 68 | 69 | 68
units on a scale | 5.46 (0.959) | 5.51 (0.956) | 3.16 (0.961)

28. Secondary Outcome: Change From Baseline in Vitality (Short Form 36-item Health Survey Domain) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 24
Time Frame: Baseline, Week 34
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 68 | 69 | 68
units on a scale | 9.88 (1.127) | 11.53 (1.123) | 5.47 (1.129)

29. Secondary Outcome: Change From Baseline in Social Functioning (Short Form 36-item Health Survey Domain) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 24
Time Frame: Baseline, Week 34
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 68
units on a scale | 8.87 (1.179) | 10.03 (1.170) | 6.42 (1.187)

30. Secondary Outcome: Change From Baseline in Role Emotional (Short Form 36-item Health Survey Domain) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 24
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 204 subjects (67 400 mg CZP, 69 200 mg CZP, 68 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 67 | 69 | 68
units on a scale | 6.86 (1.322) | 8.86 (1.313) | 5.86 (1.306)

31. Secondary Outcome: Change From Baseline in Mental Health (Short Form 36-item Health Survey Domain) at Week 34 in Patients Randomized at Week 18
Description: as for outcome 24
Time Frame: Baseline, Week 34
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 68 | 69 | 68
units on a scale | 5.38 (1.050) | 7.44 (1.042) | 4.13 (1.049)

32. Secondary Outcome: Change From Baseline in PCS (Short Form 36-item Health Survey Physical Component Summary) at Week 34 in Patients Randomized at Week 18
Description: PCS norm-based scores are calculated based upon the following 8 domain scores, Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, and range from 1 to 81, where 50 represents the normative value. A larger positive value in change from Baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 202 subjects (66 400 mg CZP, 68 200 mg CZP, 68 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 66 | 68 | 68
units on a scale | 10.54 (0.939) | 9.65 (0.928) | 5.09 (0.926)

33. Secondary Outcome: Change From Baseline in MCS (Short Form 36-item Health Survey Mental Component Summary) at Week 34 in Patients Randomized at Week 18
Description: MCS norm-based scores are calculated based upon the following 8 domain scores, Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health, and range from -9 to 82, where 50 represents the normative value. A larger positive value in change from Baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 32
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 66 | 68 | 68
units on a scale | 5.51 (1.162) | 8.59 (1.147) | 4.90 (1.143)

34. Secondary Outcome: Change From Baseline in PAAP (Patient's Assessment of Arthritis Pain) at Week 34 in Patients Randomized at Week 18
Description: Change from Baseline in Patient's Assessment of Arthritis Pain-VAS (0 to 100 mm visual analog scale, 0 being no pain and 100 being most severe pain) is computed as the value at Week 34 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 68
units on a scale | -36.41 (2.894) | -34.33 (2.869) | -17.47 (2.911)

35. Secondary Outcome: Change From Baseline in PtGADA (Patient's Global Assessment of Disease Activity) at Week 34 in Patients Randomized at Week 18
Description: Change from Baseline in Patient's Global Assessment of Disease Activity-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Week 34 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 68
units on a scale | -35.58 (2.966) | -33.07 (2.946) | -16.37 (2.987)

36. Secondary Outcome: Median Time to Loss of ACR20 (American College of Rheumatology 20% Improvement) Response After Week 18 in Patients Randomized at Week 18.
Description: ACR20 loss are subjects with <20% improvement from Baseline for tender joint count, swollen joint count, and at least 3/5 core set measures: 1) Health Assessment Questionnaire-Disability Index (HAQ-DI), 2) C-reactive Protein, 3) Patient's Assessment of Arthritis Pain-Visual Analog Scale, 4) Patient's Global Assessment of Disease Activity-Visual Analog Scale, 5) Physician's Global Assessment of Disease Activity-Visual Analog Scale at 2 consecutive visits. Subjects losing response for 2 consecutive visits are considered as having the event on the day of the visit where response was first lost.
Time Frame: Week 18 up to Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 208 subjects (69 400 mg CZP, 70 200 mg CZP, 69 placebo) are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 69
days | NA [100.0 to NA] — Because the analysis was run on the Full Analysis Set (FAS) the survival curves drop dramatically initially causing values to be non-computable. | NA [NA to NA] — Because the analysis was run on the Full Analysis Set (FAS) the survival curves drop dramatically initially causing values to be non-computable. | 98.0 [17.0 to NA] — Because the analysis was run on the Full Analysis Set (FAS) the survival curves drop dramatically initially causing values to be non-computable.

37. Other Pre Specified Outcome: Ratio From Baseline in ESR (Erythrocyte Sedimentation Rate) Level at Week 16 in All Patients
Description: Ratio is defined as the ESR value at Week 16 divided by the ESR value at Baseline. This analysis was carried out using the Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline, Week 16
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Run-in Overall
Number analyzed (Participants) | 328
Ratio | 0.6 (76.7)

38. Other Pre Specified Outcome: Ratio From Baseline in ESR (Erythrocyte Sedimentation Rate) Level at Week 34 in Patients Randomized at Week 18
Description: Ratio is defined as the ESR value at Week 34 divided by the ESR value at Baseline. This analysis was carried out using the Last Observation Carried Forward (LOCF) method with an ANCOVA model on observed log transformed data with factors treatment and log transformed Baseline CRP level. The number presented is the geometric least squares mean with it's 95% confidence interval.
Time Frame: Baseline, Week 34
Population: Of the 208 subjects in the Full Analysis Set (FAS) 205 subjects (69 400 mg CZP, 68 200 mg CZP, 68 placebo) are included in this analysis using the Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 68 | 68
Ratio | 0.56 [0.48 to 0.65] | 0.62 [0.53 to 0.72] | 0.84 [0.71 to 0.98]

39. Other Pre Specified Outcome: Change From Baseline in PhGADA (Physician's Global Assessment of Disease Activity) at Week 34 in Patients Randomized at Week 18
Description: Change from Baseline in Physician's Global Assessment of Disease Activity-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Week 34 minus the Baseline value. A negative value in change from Baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 67
units on a scale | -44.62 (2.428) | -40.24 (2.427) | -25.97 (2.476)

40. Other Pre Specified Outcome: Change From Baseline in TJC (Tender Joint Count) at Week 34 in Patients Randomized at Week 18
Description: Change from Baseline in Tender Joint Count is computed as the value at Week 34 minus the Baseline value (28 joints were assessed at each visit). A negative value in change from Baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 68
Joints | -11.81 (0.702) | -11.33 (0.692) | -7.16 (0.707)

41. Other Pre Specified Outcome: Change From Baseline in SJC (Swollen Joint Count) at Week 34 in Patients Randomized at Week 18
Description: Change from Baseline in Swollen Joint Count is computed as the value at Week 34 minus the Baseline value (28 joints were assessed at each visit). A negative value in change from Baseline indicates an improvement. This analysis was carried out using an ANCOVA model on Last Observation Carried Forward (LOCF) data with factors treatment and Baseline score.
Time Frame: Baseline, Week 34
Population: as for outcome 21
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Number analyzed (Participants) | 69 | 70 | 68
Joints | -9.29 (0.542) | -8.37 (0.540) | -5.41 (0.547)

ADVERSE EVENTS:
Time Frame: The first column represents Adverse Event (AE) reporting for the 16-Week run-in period. The last three columns represents AE reporting for the 18-Week double-blind period.
Description: Of the 209 randomized participants, 208 are in the Full Analysis Set (FAS), as 1 subject was randomized but did not receive treatment during the Double-Blind (DB) period.
Arm/Group | Run-in Overall | Certolizumab Pegol 400 mg and Placebo + Methotrexate | Certolizumab Pegol 200 mg and Placebo + Methotrexate | Placebo + Methotrexate
Serious Adverse Events (participants affected / at risk) | 18/333 | 2/69 | 5/70 | 0/69
Other Adverse Events (participants affected / at risk) | 80/333 | 20/69 | 12/70 | 27/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Overall (N=333) | Certolizumab Pegol 400 mg and Placebo + Methotrexate (N=69) | Certolizumab Pegol 200 mg and Placebo + Methotrexate (N=70) | Placebo + Methotrexate (N=69)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic peritoneal adhesions (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Overall (N=333) | Certolizumab Pegol 400 mg and Placebo + Methotrexate (N=69) | Certolizumab Pegol 200 mg and Placebo + Methotrexate (N=70) | Placebo + Methotrexate (N=69)
Nasopharyngitis (Infections and infestations) | 7 (7) | 1 (1) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 42 (46) | 8 (8) | 5 (6) | 10 (11)
Urinary tract infection (Infections and infestations) | 27 (31) | 6 (6) | 5 (5) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 5 (5) | 1 (1) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 2 (2) | 1 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.